CLINICAL TRIAL: NCT03014297
Title: A Phase 1 Study of Fosbretabulin in Combination With Everolimus in Neuroendocrine Tumors (Grades 1-3) That Have Progressed After at Least One Prior Regimen for Metastatic Disease
Brief Title: Fosbretabulin With Everolimus in Neuroendocrine Tumors With Progression
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Part I completed. Part 2 will not be done due to sponsor decision.
Sponsor: Lowell Anthony, MD (Other)
Responsible Party: Sponsor-Investigator, Lowell Anthony, MD, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16-GI-99-PMC
Record Dates: First submitted 2016-12-21; First posted 2017-01-09 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Neuroendocrine Tumors; Everolimus
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Everolimus; fosbretabulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- everolimus + fosbretabulin (Experimental): everolimus + fosbretabulin
  Interventions: Drug: everolimus; Drug: fosbretabulin

INTERVENTIONS:
Drug: everolimus — everolimus
Drug: fosbretabulin — fosbretabulin

SUMMARY:
This is a single center, open label, phase I study involving grade I-III gastroenteropancreatic neuroendocrine tumors, consisting of a dose escalation Part A followed by an expansion cohort Part B. On Part A Patients will be treated with daily oral everolimus. Fosbretabulin will be administered IV either q3 weekly or q weekly based on PO CRM cohort. Part B: Once the investigators have established an MTD in Part A, the investigators will be treating 15 more patients at that dose combination. The primary and secondary objectives of the expansion cohort will be similar to Part A of the study, i.e., to establish a safety profile of the experimental drug combination and to collect and assess efficacy data. Patients will be treated with concurrent everolimus and fosbretabulin for 12 weeks.

DETAILED DESCRIPTION:
A variety of treatment options are available for NETs with carcinoid syndrome including surgical and medical therapies. Most subjects require somatostatin analogs to control the symptoms of carcinoid syndrome. Subjects who no longer respond to somatostatin and other liver-directed therapies, who experience progression of disease and increasing symptoms have limited options, including participation in a clinical trial. Recently everolimus and sunitinib have been approved for the treatment of subjects with progressive locally advanced or metastatic neuroendocrine tumors. Based on the preclinical data in models of NETs and the clinical activity seen in NETS and other tumor types that have existing tumor vascculature, this study will examine the effectiveness of fosbretabulin given in combination with everolimus in subjects with GI-NETs and PNETs.The vasoconstrictive effect of fosbretabulin is potent, though short-lived (4-8 hours), with no cumulative adverse effect. Everolimus inhibits angiogenesis, slows tumor growth and has a prolonged half-life (30 hours). Combining these two agents with distinctly different mechanisms of action may improve tumor control without additional toxicities, and has the potential of reducing drug resistance.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed neuroendocrine tumor (grades 1-3) that is metastatic or unresectable, and for which standard curative or palliative measures do not exist or are no longer effective.
* Prior treatment with fosbretabulin is allowed, if not given in combination with everolimus.
* Prior treatment with everolimus is allowed, if the patient was able to tolerate 10 mg daily everolimus with acceptable side effects, and if everolimus was not given in combination with fosbretabulin. A 1 week washout period will be required if patient was previously on everolimus.
* Age ≥18 years.
* ECOG performance status ≤2.
* Life expectancy greater than 6 months.
* Progressive disease based on radiological imaging within 12 months. RECIST 1.1 would be used to assess measurable disease burden.
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥1,000/mcL
  * platelets ≥75,000/mcL
  * total bilirubin ≤2.5 × institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of fosbretabulin and everolimus administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had prior everolimus but were not able to tolerate a 10 mg daily dose.
* Prior chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Child Pugh Class B or greater hepatic dysfunction.
* Patients who are receiving any other investigational agents.
* Patients with known brain metastases because of their poor prognosis and likelihood to develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to fosbretabulin
* Uncontrolled hypertension (HTN); sustained blood pressure (BP) greater than 150/100 mmHg
* Must not have had any unstable angina or myocardial infarction within 4 months prior to enrollment to treatment, NYHA Class III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless subject has a pacemaker.
* Must not have any evidence of other clinically active cancer and have no history of prior malignancy within the past 3 years with the exception of: a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less and with stable prostatespecific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival for the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal glands or pancreas.
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Pregnant women are excluded from this study because everolimus and fosbretabulin have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events to nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued if the mother is treated with everolimus and fosbretabulin.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with everolimus and fosbretabulin. In addition, these patients are at increased risk of lethal infections when treated with marrowsuppressive therapy. Appropriate studies will be initiated for patients receiving combination antiretroviral therapy when indicated.
* History of prior cerebrovascular event, (including transient ischemic attack) within 6 months of start of screening.
* Current thrombotic or hemorrhagic disorder/event or history of prior event within 6 months of start of Screening
* Corrected QT interval ([QTc] Fridericia) > 480 ms
* Significant vascular disease or recent peripheral arterial thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 12 weeks
  To establish the maximum tolerated dose of the combination of everolimus plus fosbretabulin in neuroendocrine tumors (Grades 1-3) who have progressed after at least one prior regimen for metastatic disease.

SECONDARY OUTCOMES:
Incidence of Toxicities | 12 weeks
  Incidence of patients reporting at least one adverse event per NCI CTCAE v4.0
Anti-tumor activity | 12 weeks
  Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes.

CONTACTS AND LOCATIONS:
Overall Officials: Lowell Anthony, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No